CLINICAL TRIAL: NCT00135499
Title: Randomized Study of ACVBP Plus Rituximab Versus CHOP Plus Rituximab in Non Previously Treated Patients Aged From 60 to 65 Years With Diffuse Large B-Cell Lymphoma
Brief Title: R-ACVBP Versus R-CHOP in Patients Aged 60-65 With Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment too low
Sponsor: Lymphoma Study Association (Other)
Collaborators: Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNH01-5B
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Large-Cell, Diffuse
Keywords: Lymphoma; chemotherapy; rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Rituximab; Doxorubicin; Cyclophosphamide; Vindesine; Bleomycin; Prednisone; Vincristine

ARMS (2):
- R-ACVBP (Experimental): Rituximab, Doxorubicin, Cyclophosphamide, Vindesine, Bleomycin, Prednisone
  Interventions: Drug: Rituximab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vindesine; Drug: Bleomycin; Drug: Prednisone
- R-CHOP (Active Comparator): Rituximab, Doxorubicin, Cyclophosphamide, Vincristine, Prednisone
  Interventions: Drug: Rituximab; Drug: Prednisone; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vincristine

INTERVENTIONS:
Drug: Rituximab — 375 mg/m², D1, 4 cycles
Drug: Doxorubicin — 75 mg/m², D1, 4 cycles
  Arms: R-ACVBP
Drug: Cyclophosphamide — 1200 mg/m², D1, 4 cycles
  Arms: R-ACVBP
Drug: Vindesine — 2 mg/m², D1, D5, 4 cycles
  Arms: R-ACVBP
Drug: Bleomycin — 10 mg, D1, D5, 4 cycles
  Arms: R-ACVBP
Drug: Prednisone — 60 mg, D1-D5, 4 cycles
  Arms: R-ACVBP
Drug: Prednisone — 40 mg, D1-D5, 4 cycles
  Arms: R-CHOP
Drug: Doxorubicin — 50 mg/m², D1, 4 cycles
  Arms: R-CHOP
Drug: Cyclophosphamide — 750 mg/m², D1, 4 cycles
  Arms: R-CHOP
Drug: Vincristine — 1.4 mg/m², D1, 4 cycles
  Arms: R-CHOP

SUMMARY:
The primary objective of this study is to evaluate the efficacy of doxorubicin, cyclophosphamide, vindesine, bleomycin, and prednisone (ACVBP) plus rituximab in comparison to cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP) plus rituximab in patients aged from 60 to 65 years with non-previously treated diffuse large B-cell lymphoma as measured by the event-free survival. The goal is to obtain a 10% increase of event-free survival at 3 years.

DETAILED DESCRIPTION:
In Europe, 50% or more of new non-Hodgkin lymphoma cases occur in patients older than 60 years. More than 30% are diffuse large B-cell lymphomas (DLCL).

The CHOP chemotherapy (cyclophosphamide, doxorubicin, vincristine, prednisone) was considered as the standard treatment in this population. Nevertheless, this treatment is associated with some toxic events in elderly patients and it did does not succeed to increase the 3-year survival rate above 40%.

Two trials in patients above 60 years with DLCL cases were conducted by the GELA in the aim to improve the results of CHOP.

Protocol LNH 93-5 : The primary objective of this study was to compare CHOP to ACVBP in patients aged from 61 to 69 years with aggressive lymphoma and at least one adverse prognostic factor according to the International Prognostic Index.

Unlike the CHOP regimen, the ACVBP regimen includes a more intensive induction followed by a sequential consolidation with drugs different from those used during the induction phase, and includes a prevention of neuromeningeal relapses.

Out of 708 patients included in this study, the results have shown that:

* Complete response rate was the same in the two arms.
* Event free survival was significantly better in the ACVBP arm than the CHOP arm ( 5-year survival rate : 39% versus 29%, p=0.005).
* Overall survival was significantly better in the ACVBP arm than in the CHOP arm (the 5-year survival rate : 46% versus 38%, p=0.036).
* The ACVBP regimen was more toxic than the CHOP regimen, particularly in elderly patients (> 65 years) and in patients with a low performance status.
* Prevention of neuromeningeal relapses was necessary for these patients.

Protocol LNH 98-5, the objective of this study was to compare the association CHOP + rituximab (R-CHOP) to the CHOP regimen alone in elderly patients with non previously treated diffuse large B-cell lymphoma.

Long-term results based on data from 399 patients, with a median follow-up of 5 years were as follows :

* Complete response rate was better in the R-CHOP arm than in the CHOP arm (76% versus 61%, p<0.005).
* Significant prolongation of event-free survival (p<0.0002) and overall survival (p<0.0073) in the R-CHOP arm.
* No significant difference between the two arms in terms of toxicity. R-CHOP is now considered worldwide as the standard combination for these patients.

These conclusions invited us to propose a randomized trial comparing ACVBP + rituximab to CHOP + rituximab. The study population is limited to patients aged from 60 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diffuse large B-cell lymphoma according to the WHO classification (anti CD20 labeling)
* Aged from 60 to 65 years.
* Not previously treated.
* Ann Arbor stage II, III, IV.
* ECOG performance status 0 to 2.
* Minimum life expectancy of 3 months.
* Negative HIV, hepatitis B virus (HBV) and hepatitis C virus (HCV) serologies test 4 weeks (except after vaccination).
* Having previously signed a written informed consent.

Exclusion Criteria:

* T-cell lymphoma.
* Any history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Any serious active disease (according to the investigator's decision).
* Poor renal function (creatinine level>150micromol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils<1.5G/l or platelets<100G/l, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Adult patient under tutelage.

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2001-10-16 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2010-04-27 (Actual)

PRIMARY OUTCOMES:
event free survival | 8 years (end of study)
  percentage of patients alive with no event

SECONDARY OUTCOMES:
complete response rate | 8 years (end of study)
  percentage of patients with complete response
progression rate | 8 years (end of study)
  percentage of patients with progression
relapse rate | 8 years (end of study)
  percentage of patients with relapse
disease-free survival for complete responders | 8 years (end of study)
  percentage of patients with complete response who remain disease-free
overall survival | 8 years (end of study)
  percentage of patients alive
neuromeningeal relapse rate | 8 years (end of study)
  percentage of patients with neuromeningeal relapse
number of SAE | 8 years (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Tilly, MD, Principal Investigator — Lymphoma Study Association
Locations (8):
- Groupe d'Etude des Lymphomes de l'adulte, Yvoir, Belgium
- France (6):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif
- Schweirische Arbeitsgruppe fur klinische Krebsforschung, Lausanne, Switzerland

REFERENCES:
- [Background] Tilly H, Lepage E, Coiffier B, Blanc M, Herbrecht R, Bosly A, Attal M, Fillet G, Guettier C, Molina TJ, Gisselbrecht C, Reyes F; Groupe d'Etude des Lymphomes de l'Adulte. Intensive conventional chemotherapy (ACVBP regimen) compared with standard CHOP for poor-prognosis aggressive non-Hodgkin lymphoma. Blood. 2003 Dec 15;102(13):4284-9. doi: 10.1182/blood-2003-02-0542. Epub 2003 Aug 14. PMID 12920037
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Derived] Ghesquieres H, Larrabee BR, Haioun C, Link BK, Verney A, Slager SL, Ketterer N, Ansell SM, Delarue R, Maurer MJ, Fitoussi O, Habermann TM, Peyrade F, Dogan A, Molina TJ, Novak AJ, Tilly H, Cerhan JR, Salles G. FCGR3A/2A polymorphisms and diffuse large B-cell lymphoma outcome treated with immunochemotherapy: a meta-analysis on 1134 patients from two prospective cohorts. Hematol Oncol. 2017 Dec;35(4):447-455. doi: 10.1002/hon.2305. Epub 2016 Jun 10. PMID 27282998
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org